CLINICAL TRIAL: NCT01452880
Title: Total Intravenous Anaesthesia Using Remifentanil In Extracorporeal Shock Wave Lithotripsy (ESWL). Comparison of Two Dosages.
Brief Title: Remifentanil in Extracorporeal Shock Wave Lithotripsy
Acronym: ESWL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Cannata, medical doctor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: francesco cannata
Record Dates: First submitted 2011-10-06; First posted 2011-10-17 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Kidney Calculi
Keywords: Remifentanil; Lithotripsy; Conscious Sedation
MeSH Terms: conditions — Kidney Calculi | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Remifentanil — Remifentanil is an ultra-short-acting oppioid, which is quickly metabolized by unspecific blood and tissue esterases
Drug: Remifentanil — GROUP A (N = 114): patients assigned to this group received Remifentanil at infusion rate of 0.05 mcg / kg / min I.V. ; GROUP B (N = 114): in this group Remifentanil was administered at infusion rate of 0,1 mcg / kg / min I.V. Remifentanil was administered intravenously throughout ESWL procedure.

SUMMARY:
The purpose of this study is to compare the analgesic efficacy and side effects induced by administration of two different infusion rates of remifentanil, 0,05 mcg/ Kg/ min versus 0,1mcg/ Kg/ min, in order to determine which one is the most appropriate analgesic treatment to face extracorporeal shock wave lithotripsy.

DETAILED DESCRIPTION:
Remifentanil is an ultra-short-acting oppioid, which is quickly metabolized by unspecific blood and tissue esterases . This feature vouches for a predictable pharmacokinetics and makes this drug suitable for administration in continuous intravenous infusion in order to achieve patient conscious sedation during non-invasive surgical procedures. Remifentanil could be particularly useful in day surgery setting, thanks also to its faster elimination than other oppioids. This property ensure a swift recovery from conscious sedation, reducing the period of time during which patient remains in recovery room and decreasing also the incidence of side effects, like PONV and respiratory depression. Conscious sedation with remifentanil can provide patient comfort and cooperation during surgical procedure, since the verbal contact with the patient is kept up. Extracorporeal shock wave lithotripsy (ESWL) is a non-invasive procedure, contemplated as the first-line treatment for renal and upper ureteral stones, if stone diameter is ranged from 5 to 20 mm . It can grind calculi into fine particles, that are expelled through micturition. Although many studies have been published in regard to continuous intravenous infusion of remifentanil, a small number of them focuses on which is the most appropriate infusion rate for ESWL procedure.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of anaesthesiology) physical status between the I and class II
* Body mass index (BMI) between 18 and 30.

Exclusion Criteria:

* Patients who were unable to give informed consent or with diagnosis of depression
* Concurrent treatment with antidepressant
* Anxiolytic or with opioids or with history of abuse and dependence from these substances
* Allergy or intolerance to drugs administered in this study
* Severe cognitive deficits or psychiatric disorders
* Liver or renal impairment (aspartate aminotransferase > 40 UI/L alanine aminotransferase > 40 UI/L, creatinine > 2mg/dL)
* Abnormal values of coagulation (International normalized ratio > 1,2), platelet(< 100.000/µL), arrhythmias and / or defect of atrioventricular conduction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
VAS score | Vas score was monitored up to the end of surgery, for about forty minutes
  Before the beginning of ESWL and at the end of the treatment patient were asked to point out the intensity of pain they were feeling on an 11-points visual analog scale (VAS), ranged from 0 "no pain" to 10 "worst pain".

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cannata, medical doctor, Principal Investigator — policlinico Umberto I Sapienza University of Rome
Locations (1):
- Policlinico Umberto I, Rome, Italy/RM, Italy

REFERENCES:
- [Result] Medina HJ, Galvin EM, Dirckx M, Banwarie P, Ubben JFH, Zijlstra FJ, Klein J, Verbrugge SJC. Remifentanil as a single drug for extracorporeal shock wave lithotripsy: a comparison of infusion doses in terms of analgesic potency and side effects. Anesth Analg. 2005 Aug;101(2):365-370. doi: 10.1213/01.ANE.0000159379.54705.84. PMID 16037145
- See also: European Society of Anaesthesiology — http://www.euroanesthesia.org/